CLINICAL TRIAL: NCT02398409
Title: Telephone Assessment and Skill-Building Intervention for Informal Caregivers
Brief Title: Informal Caregivers ANSWERS-VA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: NRI 12-415
Record Dates: First submitted 2015-02-26; First posted 2015-03-25 (Estimated); Results first posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Stroke; Traumatic Brain Injury
Keywords: stroke; Injury, Brain, Traumatic; Family Caregivers; TBI (Traumatic Brain Injury); Informal Caregivers
MeSH Terms: conditions — Stroke; Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ANSWERS-VA (Experimental): 8 week telephone intervention with nurse case manager using "Acquiring New Skills While Enhancing Remaining Strengths" (ANSWERS)
  Interventions: Behavioral: ANSWERS - Acquiring New Skills While Enhancing Remaining Strengths
- Control (Other): 8 week telephone usual care with education with nurse case manager
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: ANSWERS - Acquiring New Skills While Enhancing Remaining Strengths — Randomized trial to evaluate the efficacy of the telephone intervention "Acquiring New Skills While Enhancing Remaining Strengths"in informal caregivers of Veterans with stroke and TBI.
  Arms: ANSWERS-VA
Other: Control — 8 week telephone usual care with education with nurse case manager
  Arms: Control

SUMMARY:
The purpose of this study is to determine the effectiveness of the ANSWERS- VA intervention (Acquiring New Skills While Enhancing Remaining Strengths for Veterans) while also determining it's cost effectiveness in the stroke and traumatic brain injury (TBI) populations.

DETAILED DESCRIPTION:
Background: Stroke and traumatic brain injury (TBI) are leading causes of long-term disability among Veterans and result in the need for care from informal caregivers in the home setting. There are very few evidence-based, easy-to-deliver follow-up programs to train Veterans and caregivers across multiple domains post injury. The "Acquiring New Skills While Enhancing Remaining Strengths for Veterans (ANSWERS-VA)" intervention aims to provide the Veteran and caregiver dyad with a set of practical skills that each can use in coping with and managing symptoms of a brain injury, applying a strength-based approach.

Objectives: The objectives of this study are to conduct a randomized controlled trial (RCT) to evaluate (a) the efficacy of the ANSWERS-VA dyadic intervention with Veterans who have sustained a stroke and/or TBI and their informal caregivers, and (b) estimate effect sizes for the ANSWERS-VA intervention. The ANSWERS-VA intervention will be compared with an educational intervention that will serve as an attention control group.

Specific Aim 1: To tailor the implementation of the ANSWERS-VA intervention to dyads of Veterans post stroke and/or TBI and their informal caregivers (n=10) and modify the implementation processes for the RCT.

Specific Aim 2: To test the short-term (immediately post-intervention) and long-term, sustained (12 and 24 weeks, and at 1 year) efficacy of the ANSWERS-VA intervention for improving: (a) the primary outcomes of the caregivers' quality of life and unhealthy days, and (b) the caregiver mediators of task difficulty, threat appraisal, self-efficacy for caregiving, and optimism.

Specific Aim 3: To evaluate program delivery costs for the ANSWERS-VA intervention and the educational attention control procedures, and to assess the cost-effectiveness of the ANSWERS-VA intervention in terms of noncaregiving hours and unhealthy days in caregivers of Veterans post stroke and/or TBI.

Exploratory Aim 1: To estimate the effect sizes for the ANSWERS-VA intervention for the caregiver and Veteran on the secondary outcomes of depressive symptoms, social participation, and quality of the dyadic relationship.

Methods: The investigators propose to conduct a RCT to evaluate the ANSWERS-VA intervention among Veterans with stroke or TBI and their caregivers (dyads). Veterans with stroke (N = 222) or TBI (N = 108) and their informal caregivers, who have received care at the Michael E. DeBakey Veterans Affairs Medical Center in Houston or the Richard L. Roudebush VAMC in Indianapolis, will be randomized to the ANSWERS-VA intervention or to an attention control group. Both the intervention and control procedures involve 8 telephone sessions delivered over 8 weeks, with a booster session at 12 weeks. Data collections will occur at baseline, 8 weeks (short-term intervention effect), 12 weeks (after booster), 24 weeks, and 1 year after baseline (long-term sustainability of intervention effect). Linear mixed models will be applied to the repeated-measures data to test efficacy of the program in stroke caregivers and to estimate effect sizes in TBI caregivers. An incremental cost-effectiveness ratio will be employed to address the comparative costs and outcomes for the ANSWERS-VA intervention and attention control groups.

Status: Essential modifications for this project were requested and approved via VA Central Office. Institutional Review Board approval has been obtained for these modifications in Indianapolis and in Houston. Graduate students from multiple disciplines have been hired and have received two days of onsite training specific to the ANSWERS-VA intervention and control procedures, screening, recruitment, and data collection processes. The REDCap database has been updated for the project modifications and has been further tested. The investigators are currently working with frontline providers at both sites to recruit potential participants for this RCT. Enrollment of first subject dyads began November, 2014. At this time, the investigators have completed recruitment of new dyads. We continue to complete outcomes assessments on some dyads. We plan to submit an abstract to the International Stroke Conference in January 2019.

ELIGIBILITY:
Inclusion Criteria:

* Informal caregiver of a family member or friend (Veteran) with a stroke or TBI
* Caregiver must express need or concerns in providing care
* Plans to be providing care for 1 year or longer
* Access to telephone
* Willingness to participate in 9 call from a nurse and 5 data collection calls at designated timepoints
* Veteran's stroke must be within past 3 years
* Veteran's TBI must be since 9/11/01

Exclusion Criteria:

* Caregiver or survivor age < 18 years
* Caregiver denies that survivor has had a stroke or a TBI
* Caregiver does not consider him or herself a caregiver, stating that the survivor is not impaired or is the same as before the stroke or TBI
* Caregiver has low task difficulty (OCBS task difficulty score < 16)
* Caregiver communication difficulties (e.g., hearing loss)
* Caregiver not fluent in the English language
* Caregiver with serious medical illness limiting ability to participate
* Caregiver refuses to sign a HIPAA authorization allowing the VA to store personal health information (PHI) in a location outside the VA
* Survivor residing in a nursing home or long-term care facility
* Survivor or caregiver has a terminal illness (e.g., cancer, end of life condition with decreased life expectancy, renal failure requiring dialysis)
* Survivor or caregiver history of hospitalization for alcohol or drug abuse
* Survivor or caregiver history of Alzheimer's, dementia, suicidal tendencies, severe untreated depression or manic depressive disorder, or schizophrenia.
* Survivor or caregiver pregnancy
* Survivor or caregiver is a prisoner or on house arrest
* Survivor had a Transient Ischemic Attack (rather than a hemorrhagic or ischemic stroke)
* Survivor had a stroke more than 3 years ago

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2014-11-03 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2019-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Virginia (Ginger) S. Wilder, PhD MSN RN, Principal Investigator — Richard L. Roudebush VA Medical Center, Indianapolis, IN
Locations (2):
- United States (2):
  - Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Crocker TF, Brown L, Lam N, Wray F, Knapp P, Forster A. Information provision for stroke survivors and their carers. Cochrane Database Syst Rev. 2021 Nov 23;11(11):CD001919. doi: 10.1002/14651858.CD001919.pub4. PMID 34813082

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The number of recruited participants (143) is slightly different from the number of participants represented in the flow diagram (137) due to the fact there were 6 participants after recruitment and informed consent we were not able to reach them for data collection.
Pre-assignment Details: Veterans and Caregiver were enrolled as dyads. "Participants" refers to the Dyads.
Groups:
- ANSWERS-VA: 8 week telephone intervention with nurse case manager using "Acquiring New Skills While Enhancing Remaining Strengths" (ANSWERS)
  ANSWERS - Acquiring New Skills While Enhancing Remaining Strengths: Randomized trial to evaluate the efficacy of the telephone intervention "Acquiring New Skills While Enhancing Remaining Strengths"in informal caregivers of Veterans with stroke and Traumatic Brain Injury (TBI).
Period: Overall Study
Arm/Group | ANSWERS-VA | Control
Started | 69 | 68
Completed | 67 | 63
Not Completed | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ANSWERS-VA | Control | Total
Number analyzed (Participants) | 67 | 63 | 130
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 57 | 50 | 107
  >=65 years | 10 | 13 | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 57 | 118
  Male | 6 | 6 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Caregiver's Depressive Symptoms by Patient Health Questionnaire (PHQ9) Scale
Description: Depression scores are measured with the PHQ9 scale. Scores can range from 0 to 27, with higher scores indicating higher levels of depression.
Time Frame: Baseline, Week 12, 6 months and 1 year
Population: Not change data. One Intervention Caregiver and one Control Caregiver did not complete the PHQ9. Those data are missing.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ANSWERS-VA | Control
Number analyzed (Participants) | 66 | 62
score on a scale
  Baseline | .56 (.53) | .68 (.61)
  Week 12: number analyzed (Participants) | 15 | 29
  Week 12 | .41 (.45) | .62 (.59)
  6 Months: number analyzed (Participants) | 14 | 26
  6 Months | .20 (.25) | .57 (.56)
  1 Year: number analyzed (Participants) | 16 | 22
  1 Year | .47 (.66) | .43 (.49)
Statistical Analysis 1: Comparison: ANSWERS-VA; 12 weeks compared to Baseline (BL); Test type: Superiority; p = .8407, Mixed Models Analysis — Adjusting for the covariates of diagnosis and baseline mean value in caregivers' depression; Mean Difference (Net) = .016, Standard Error of Mean .117
Statistical Analysis 2: Comparison: ANSWERS-VA; At 6 months compared to BL; Test type: Superiority; p = .0150, Mixed Models Analysis — Adjusting for the covariates of diagnosis and baseline mean value in caregivers' depression; Median Difference (Net) = .201, Standard Error of Mean .120
Statistical Analysis 3: Comparison: ANSWERS-VA; 1 year compared BL; Test type: Superiority; p = .8373, Mixed Models Analysis — adjusting for the covariates of diagnosis and baseline mean value in caregivers' depression; Median Difference (Net) = .114, Standard Error of Mean .188

2. Primary Outcome: Mediators of Caregiver's Task Difficulty
Description: Task difficulty is measured with the Oberst Caregiving Burden Scale. Scores on a Likert scale can range from 1 to 5 with higher scores indicating higher levels of burden.
Time Frame: Baseline, Week 12, 6 months and 1 year
Population: Not change data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ANSWERS-VA | Control
Number analyzed (Participants) | 67 | 63
score on a scale
  Baseline | 1.99 (.77) | 1.83 (.68)
  12 Week: number analyzed (Participants) | 15 | 29
  12 Week | 1.73 (.70) | 1.73 (.61)
  6 Months: number analyzed (Participants) | 14 | 26
  6 Months | 1.70 (.64) | 1.63 (.57)
  1 Year: number analyzed (Participants) | 16 | 22
  1 Year | 1.78 (.62) | 1.66 (.79)
Statistical Analysis 1: Comparison: ANSWERS-VA; 12 weeks compared to BL; Test type: Superiority; p = .6445, Mixed Models Analysis — adjusting for the covariates of diagnosis and baseline mean value in caregivers' depression; Median Difference (Net) = .016, Standard Error of Mean .173
Statistical Analysis 2: Comparison: ANSWERS-VA; 6 months compared to BL; Test type: Superiority; p = .5247, Mixed Models Analysis — adjusting for the covariates of diagnosis and baseline mean value in caregivers' depression; Median Difference (Net) = .033, Standard Error of Mean .158
Statistical Analysis 3: Comparison: ANSWERS-VA; 1 year compared to BL; Test type: Superiority; p = .9974, Mixed Models Analysis — adjusting for the covariates of diagnosis and baseline mean value in caregivers' depression; Median Difference (Net) = .1224, Standard Error of Mean .187

3. Primary Outcome: Mediators of Caregiver's Optimism Scale
Description: Optimism is measured with the Life Orientation Test-Revised Scale. Scores can range from 0 to 40 with higher scores indicating more optimism.
Time Frame: Baseline, Week 12, 6 months and 1 year
Population: Not change data. One Control Caregiver did not complete the Life Orientation Test-Revised Scale. Those data are missing.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ANSWERS-VA | Control
Number analyzed (Participants) | 67 | 62
score on a scale
  Baseline | 2.29 (.35) | 2.33 (.39)
  12 Week: number analyzed (Participants) | 15 | 29
  12 Week | 2.19 (.40) | 2.29 (.27)
  6 Months: number analyzed (Participants) | 14 | 26
  6 Months | 2.31 (.34) | 2.29 (.31)
  1 Year: number analyzed (Participants) | 16 | 22
  1 Year | 2.25 (.27) | 2.28 (.37)
Statistical Analysis 1: Comparison: ANSWERS-VA; 12 weeks compared to BL; Test type: Superiority; p = .1918, Mixed Models Analysis — adjusting for the covariates of diagnosis and baseline mean value in caregivers' depression; Median Difference (Net) = .054, Standard Error of Mean .087
Statistical Analysis 2: Comparison: ANSWERS-VA; 6 months compared to BL; Test type: Superiority; p = .9212, Mixed Models Analysis — adjusting for the covariates of diagnosis and baseline mean value in caregivers' depression; Median Difference (Net) = .046, Standard Error of Mean .078
Statistical Analysis 3: Comparison: ANSWERS-VA; 1 year compared to BL; Test type: Superiority; p = .2358, Mixed Models Analysis — adjusting for the covariates of diagnosis and baseline mean value in caregivers' depression; Median Difference (Net) = .026, Standard Error of Mean .083

4. Primary Outcome: Mediators of Caregiver's Threat Appraisal Scale
Description: Threat appraisal is measured with the Appraisal of Caregiving Scale: Threat Subscale. Scores on a Likert scale can range from 1 to 5 with higher scores indicating less belief, feelings and ability to take care of a loved one with stroke or brain injury in the future.
Time Frame: Baseline, Week 12, 6 months and 1 year
Population: Not change data. One Control Caregivers did not complete the Threat Subscale. Those data are missing.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ANSWERS-VA | Control
Number analyzed (Participants) | 67 | 62
score on a scale
  Baseline | 2.73 (.86) | 2.66 (.78)
  12 Week: number analyzed (Participants) | 15 | 29
  12 Week | 2.56 (.83) | 2.49 (.68)
  6 Months: number analyzed (Participants) | 14 | 26
  6 Months | 2.38 (.95) | 2.69 (.67)
  1 Year: number analyzed (Participants) | 16 | 22
  1 Year | 2.58 (1.0) | 2.44 (.61)
Statistical Analysis 1: Comparison: ANSWERS-VA; 12 weeks compared to BL; Test type: Superiority — adjusting for the covariates of diagnosis and baseline mean value in caregivers' depression; p = .1107, Mixed Models Analysis; Median Difference (Net) = .008, Standard Error of Mean .168
Statistical Analysis 2: Comparison: ANSWERS-VA; 6 months compared to BL; Test type: Superiority — adjusting for the covariates of diagnosis and baseline mean value in caregivers' depression; p = .0562, Mixed Models Analysis; Median Difference (Net) = .251, Standard Error of Mean .211
Statistical Analysis 3: Comparison: ANSWERS-VA; 1 year compared to BL; Test type: Superiority; p = .8579, Mixed Models Analysis — adjusting for the covariates of diagnosis and baseline mean value in caregivers' depression; Median Difference (Net) = .226, Standard Error of Mean .218

ADVERSE EVENTS:
Time Frame: Baseline to 12 month follow up.
Arm/Group | ANSWERS-VA | Control
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/63
Other Adverse Events (participants affected / at risk) | 2/67 | 0/63
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ANSWERS-VA (N=67) | Control (N=63)
Adverse Event (Cardiac disorders) | 1 (1) | 0 (0) — Participant presented to local Emergency Department with chest pains. Diagnosed with A-fib, released to home and told to follow up with Primary Care Physician.
adverse event (Cardiac disorders) | 1 (1) | 0 (0) — Participant reported she had a minor heart attack in September. This was reported to research personnel at an outcomes calls. Hospitalized overnight at local hospital and released to home.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-09-15): https://cdn.clinicaltrials.gov/large-docs/09/NCT02398409/Prot_SAP_000.pdf
  • Informed Consent Form (2016-03-24): https://cdn.clinicaltrials.gov/large-docs/09/NCT02398409/ICF_001.pdf